CLINICAL TRIAL: NCT02922478
Title: Role of Comorbidities in Chronic Heart Failure (RoC-HF) Study
Brief Title: Role of Comorbidities in Chronic Heart Failure Study
Acronym: RoC-HF
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Dirk von Lewinski, Clinical Professor, Medical University of Graz
Other Study IDs: 28-476 ex 15/16
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure; Comorbidity; Osteoporosis; Pulse Wave Analysis; Blood Pressure Monitoring, Ambulatory; Osteoporotic Fractures
MeSH Terms: conditions — Heart Failure; Osteoporosis; Osteoporotic Fractures | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — EDTA plasma, serum and buffy coat will be stored at -80 °C for later determination of biomarkers and DNA sequencing.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: X-ray of the spine — Every participant will undergo X-ray of the spine so that vertebral fractures can be quantified using the Genant score.
Procedure: Ambulatory blood pressure monitoring (ABPM) — ABPM will be performed using the brachial, oscillometric, automated self-measurement mobil-O-Graph device (I.E.M. GmbH, Stolberg, Germany) with integrated ARCSolver®-Software (Austrian Institute of Technology Wien).
Radiation: Dual X-ray absorptiometry — Individual bone mineral density and T-Score will be determined by X-ray absorptiometry.
Procedure: Non-invasive procedures — Other non-invasive study procedures include structured patient interview, sampling of blood, buffy coat and spot urine (including biobanking), electrocardiogram, pulse wave velocity and analysis, transthoracic echocardiography, 4-meter gait speed test, hand grip test, questionnaires

SUMMARY:
This study aims to create a database of patients with stable and chronic heart failure with comprehensive assessment of bone, skeletal and vascular status. RoC-HF will facilitate cross-sectional and, eventually, longitudinal mechanistic epidemiological analyses to disentangle the role of the bone- vascular axis in chronic heart failure. Blood and urine samples will be stored to facilitate future biomarker analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18
2. NYHA (New York Heart Association) class II-IV symptoms
3. Left ventricular ejection fraction < 50% at Visit 1.
4. Treatment according to current Heart Failure Guidelines of the European Society of Cardiology
5. Willingness and ability to provide signed informed consent form (ICF) prior to participation in any study-related procedures
6. Previous diagnosis of heart failure with reduced ejection fraction defined as symptomatic left ventricular ejection < 40% requiring optimization of heart failure therapy

Exclusion Criteria:

1. Unplanned hospitalization within 1 month prior to the Baseline Visit.
2. Discontinuation or initiation of a pharmacologic or device treatment for HFrEF within 1 month prior to the baseline visit.
3. Coronary or peripheral revascularization procedures, valvular procedures, OR any major surgical procedure within 3 months prior to the Screening Visit.
4. Acute coronary syndrome (ACS), stroke or transient ischemic attack (TIA) within 3 months prior to the Screening Visit.
5. Any acute illness
6. Disease reducing life expectancy to < 1 year, except HFrEF
7. Recipient of any organ transplant
8. Primary significant valve disease (at least moderate to severe valve disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable patients with chronic heart failure
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of osteoporosis in chronic heart failure | 1 day
Prevalence of vertebral fractures in chronic heart failure | 1 day

SECONDARY OUTCOMES:
Peripheral and central pulse wave velocity | 24 hours
24-hours systolic and diastolic blood pressure | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Verheyen, MD, Principal Investigator — Medical University of Graz; Klemens Ablasser, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02922478/Prot_SAP_000.pdf